CLINICAL TRIAL: NCT00505960
Title: Diabetes Care for Korean Americans
Brief Title: Culturally Tailored Behavioral Diabetes Care Intervention for Korean Americans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Miyong T. Kim, The Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R34DK071957 (NIH)
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Behavioral: Diabetes Care for Korean Americans

INTERVENTIONS:
Behavioral: Diabetes Care for Korean Americans — Intervention group participants receive a 6-week in-class education offered by trained nurses, followed by home glucose monitoring with monthly nurse telephone counseling.

SUMMARY:
The purpose of this study is to assess the feasibility and efficacy of a culturally-tailored, comprehensive behavioral intervention program specially designed for linguistically challenged ethnic minority immigrant populations (Korean Americans) with type 2 DM.

DETAILED DESCRIPTION:
Korean American immigrants (KAI), one of the most underserved and understudied minority populations in the U.S., suffer from diabetes, which goes under-diagnosed, inadequately treated and has a potential to result in costly and tragic consequences. Language barriers, the lack of self-confidence, and diminished social support that accompany the acculturation process prevent KAI from improving their health-seeking behaviors. Our previous research has indicated that overwhelming numbers of KAI suffer not only from uncontrolled hyperglycemia but also from a loss of self-confidence and social isolation because of language and cultural barriers. They are in urgent need of an intervention to assist them in their efforts to achieve better glycemic control and restore their self-confidence in diabetes and health management so that they are able to adjust successfully in this new environment. Therefore, The purpose of this study is to assess the feasibility and efficacy of a culturally-tailored, comprehensive behavioral intervention program specially designed for linguistically challenged KAIs with type 2 DM.

This pilot project will test the hypothesis: Compared to KAI in the control group, KAI with type 2 DM who receive a comprehensive DM management intervention through structured psycho-behavioral education, home glucose monitoring with a telephone transmission system, and interaction with a bilingual nurse case manager will show: (1) a greater level of glucose control; and (2) a greater level of self-help skills including knowledge related to glucose control, problem-solving skills, heightened confidence and mood/affect, adherence to treatment recommendations, and quality of life. An additional outcome will be to measure and obtain an ideal BP as the proposed intervention focuses on management of multiple risk factors with which many KA DM patients often struggle.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as a first generation Korean American
* Age 30 years or older
* Resides in Washington-Baltimore area
* Expresses willingness to participate in all aspects of the study over its full course
* Written consent to participate in the screening/eligibility visit
* Self-identified with DM and HbA1c >= 8% within 6 months of screening
* Written consent to participate in the clinical trial: agreeing to participate in study data collection procedures, receiving DM self -help education, using HGMT, and permitting contact with their own medical care provider.

Exclusion Criteria:

* Unable to give informed consent
* Physical or mental health conditions that could limit active participation in the study (e.g., blindness in both eyes, severe immobility, psychiatric diseases)
* Hematological condition that would affect A1C assay, e.g., hemolytic anemia, sickle cell anemia.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | 30 Weeks
  The primary outcome varialbe is hemoglobin A1c level of the study participants to assess the status of blood gluocse management and control during previous 2-3 months.

SECONDARY OUTCOMES:
BP control | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miyong T Kim, PhD, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Korean Resource Center, Ellicott City, Maryland, United States

REFERENCES:
- [Background] Song HJ, Han HR, Lee JE, Kim J, Kim KB, Nguyen T, Kim MT. Translating current dietary guidelines into a culturally tailored nutrition education program for Korean American immigrants with type 2 diabetes. Diabetes Educ. 2010 Sep-Oct;36(5):752-61. doi: 10.1177/0145721710376328. Epub 2010 Jul 22. PMID 20651099
- [Result] Kim MT, Han HR, Song HJ, Lee JE, Kim J, Ryu JP, Kim KB. A community-based, culturally tailored behavioral intervention for Korean Americans with type 2 diabetes. Diabetes Educ. 2009 Nov-Dec;35(6):986-94. doi: 10.1177/0145721709345774. PMID 19934458
- [Derived] Nam S, Han HR, Song HJ, Song Y, Kim KB, Kim MT. Utility of a point-of-care device in recruiting ethnic minorities for diabetes research with community partners. J Health Care Poor Underserved. 2011 Nov;22(4):1253-63. doi: 10.1353/hpu.2011.0117. PMID 22080707